CLINICAL TRIAL: NCT07014527
Title: Assessment of the Accuracy of Full Digital Workflow in Patient Specific Submerged Subperiosteal Implants: A Case Series Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Shawky, Assistant lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMFS 2025
Record Dates: First submitted 2025-05-25; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-01

CONDITIONS: Edentulous Alveolar Ridge Atrophy; ATROPHYC EDENTULOUS JAW; Edentulous Maxilla; Edentulous Alveolar Ridge In Mandible

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computer guided custom made subperiosteal implant treatment (Experimental): Patients will receive a patient specific custom made subperiosteal implant and the accuracy will be assessed
  Interventions: Procedure: Patient specific subperiosteal implants

INTERVENTIONS:
Procedure: Patient specific subperiosteal implants — Patient specific subperiosteal implants

SUMMARY:
custom made subperiosteal implants will be designed using the patients' CT data and will be inserted with the help of a surgical guide and loaded by a screw retained full arch prosthesis. accuracy will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Adults patients with severely atrophic alveolar ridges in both maxilla and mandible.

Exclusion Criteria:

* Alveolar bone dimensions that can allow for root form implant placement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Accuracy | immediately postoperative
  accuracy of the position of patient specific subperiosteal implants by superimposition of immediately postoperative CT over the preoperative plan and taking linear measurements (in millimeters)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request from the authors